# STATISTICAL ANALYSIS PLAN

### **Trial Title:**

Two-site laboratory-based diagnostic accuracy and feasibility study of the Xpert MTB/XDR assay for detection of isoniazid, fluoroquinolone, ethionamide and second-line injectable anti-tuberculosis drug resistance

#### Short title:

TB-CAPT MTB/XDR Study

Version: 1.2

Date: 28 March 2021

Funder: EDCTP

Sponsor Name: FIND Disease Programme: TB

Protocol number: 1.0

Study Statistician: Stefano Ongarello Consultant on sample size calculation: Thomas Keller (Acomed Statistik)



FIND

Campus Biotech

Chemin des Mines 9

1202 Geneva

Switzerland

T: +41 (0)22 710 05 90

F: +41 (0)22 710 05 99

| Name and Function | Date | Signature |
|---|---|---|
| | DD/MM/YYYY | |
| SAP Author | | |
| Chad Centner | | |
| Pathologist | | |
| National Health Laboratory<br>Service | 28-03-2021 | farman |
| University of Cape Town | | |
| Supervisor of SAP author | | |
| Helen Cox | 28 March 2021 | Heler Com |
| Trial Manager | | |
| Adam Penn-Nicholson | 31 March 2021 | The |
| Head of Data Services and Biobanking (if not author) | | |
| Stefano Ongarello | 31MAR2021 | APQ16 |

#### **CONFIDENTIALITY STATEMENT:**

The information contained in this document is confidential and the property of FIND (or under its control). The information may not (in full or in part) be transmitted, reproduced, published, or disclosed to others without prior written authorization from FIND, except where necessary to obtain informed consent from those who will participate in the study.

#### Table of contents Introduction ......5 1.1 Description of the study .......5 1.2 Timing of the analysis ......5 Statistical hypotheses and methods ......5 2 2.1 Primary endpoints......5 2.2 Secondary endpoints ......6 Trial population and analysis datasets......7 3.1 Criteria for eligibility, recruitment, withdrawal and follow-up ......8 32 Analysis datasets......8 Description of statistical methods .......8 General approach ......  4.1 4.2 Analysis of the primary outcome(s) ......9 4.3 Analysis of the secondary outcome(s)......  5 6 Planned interim analyses......11 7 Additional sub-group analyses......11 8 Multiple comparisons/multiplicity adjustments ......11 Exploratory analyses......11 9 10 Sample size......11 11 Minimization of error and bias ......14 11.1 12 13 14 15 Appendix .....  16

### 1 Introduction

This document describes the statistical analysis plan for the following project: "Two-site laboratory-based diagnostic accuracy and feasibility study of the Xpert MTB/XDR assay for detection of isoniazid, fluoroquinolone, ethionamide and second-line injectable anti-tuberculosis drug resistance."

### 1.1 Description of the study

The study aims to evaluate the Xpert MTB/XDR cartridge by estimating the diagnostic accuracy of the assay for the detection of resistance to isoniazid, fluoroquinolones, ethionamide and second-line injectable anti-tuberculosis drugs in clinical specimens positive for rifampicin-resistant *Mycobacterium tuberculosis* (*Mtb*) by Xpert MTB/RIF Ultra, using a composite reference standard. The composite reference standard comprises phenotypic susceptibility testing and whole genome sequencing (WGS) performed on culture isolates.

Secondary aims of the project are to estimate the diagnostic accuracy of Xpert MTB/XDR for detection of resistance to isoniazid, fluoroquinolones and second-line injectable anti-tuberculosis drugs compared to each method alone. Further secondary aims are to compare the diagnostic accuracy of the MTB/XDR assay to that of standard of care (SOC) testing, as well as compare the turnaround time (time-to-result) of Xpert MTB/XDR versus SOC. SOC at the two sites includes direct and indirect (culture-based) line probes assays (LPA)s.

Additionally, the study will investigate the feasibility of performing Xpert MTB/XDR on residual SR-sputum mix of rifampicin-resistant respiratory samples leftover from the Xpert MTB/RIF Ultra, under routine conditions.

## 1.2 Timing of the analysis

The final analysis will be conducted once all results are available (i.e. enrolment is complete and all phenotypic DST and genotypic testing results have been returned). All objectives will be analysed together at this time.

## 2 Statistical hypotheses and methods

## 2.1 Primary endpoints

- The primary endpoint is the estimate of sensitivity and specificity of Xpert MTB/XDR assay vs. the composite reference standard for detection of resistance to:
  - a. Isoniazid

- b. Fluoroquinolones
- c. Ethionamide
- d. Second-line injectable anti-tuberculosis drugs

### 2.2 Secondary endpoints

- 1. Point estimated of sensitivity and specificity of Xpert MTB/XDR for detection of resistance to:
  - a. Isoniazid
  - b. Fluoroguinolones
  - c. Second-line injectable anti-tuberculosis drugs

compared to phenotypic anti-tuberculosis drug susceptibility testing and WGS separately

- 2. Point estimates of sensitivity and specificity of Xpert MTB/XDR vs. WGS for detection of mutations in the following gene targets:
  - a. inhA promoter
  - b. katG
  - c. gyrA
  - d. gyrB
  - e. eis
  - f. rrs
- 3. Point estimates of sensitivity and specificity of Xpert MTB/XDR compared to that of SOC testing against the composite reference standard for detection of resistance to:
  - a. Isoniazid
  - b. Fluoroguinolones
  - c. Second-line injectable anti-tuberculosis drugs
- 4. Estimate of the proportion of participants for whom valid test results become available based on:
  - a. Xpert MTB/XDR
  - b. SOC testing:
    - i. LPAs performed directly on specimen ("direct")
    - ii. LPAs performed on culture isolates ("indirect")
- 5. Estimate of the median time-to-result (time in hours from sample receipt to finalised result):
  - a. Separately for each drug class, and comparing:
    - i. Xpert MTB/XDR
    - ii. SOC testing:

- 1. Direct LPAs
- 2. Indirect LPAs

#### 6. Feasibility endpoints:

- a. Estimate of the proportion of participants with sufficient residual SR-sputum mix (≥2 ml) available to perform Xpert MTB/XDR
- Median period between preparation of SR-sputum mix and start of Xpert MTB/XDR test
- c. Estimate of the proportion of specimens with non-determinate MTB/XDR results:
  - i. Combined for all
  - ii. Separately for each drug class
  - iii. Separately for each target gene
  - iv. Comparing specimens stored according to manufacturer recommendations (at 2-8°C for ≤4 hours or 25-35°C for ≤2.5 hours) and those exceeding those limits for operational reasons
  - v. By subgroup:
    - 1. Sufficient specimen (yes/no)
    - 2. Smear status
    - 3. Age group

### 7. Exploratory endpoints:

- a. Point estimates of sensitivity and specificity of Xpert MTB/XDR assay for detection of resistance to each anti-tuberculosis drug class by subgroup:
  - i. Sufficient specimen (yes/no)
  - ii. Smear status
  - iii. Age group
- Point estimates of sensitivity and specificity of Xpert MTB/XDR assay for detection of resistance to each anti-tuberculosis drug class by rifampicin susceptibility result concordance between Xpert MTB/RIF Ultra and LPA
- c. Estimates of the agreement (kappa statistic) between Xpert MTB/XDR and WGS for the detection of heteroresistance for each antituberculosis drug class
- d. Description of discordance between phenotypic testing and WGS
- e. Description of discordance between testing methodologies by presence of heteroresistance

## 3 Trial population and analysis datasets

### 3.1 Criteria for eligibility, recruitment, withdrawal and follow-up

#### Inclusion:

 Mtb-positive, rifampicin-resistant respiratory specimen identified on Xpert MTB/RIF Ultra

#### **Exclusion:**

- Residual SR-sputum mix not retained or not found
- Patient previously included in the study

Exclusion for diagnostic accuracy and time-to-result endpoints:

- Insufficient residual SR-sputum mix remaining for Xpert MTB/XDR (<2 ml)</li>
- Xpert MTB/XDR unsuccessful
- No second / follow-up specimen received
- Second / follow-up specimen culture-negative, contaminated or not available
- Reference standard uninterpretable (phenotyping or WGS)
  - Where phenotypic susceptibility testing results are uninterpretable, specimens will still be included in WGS comparison
  - Where WGS results are uninterpretable, specimens will still be included in phenotypic susceptibility testing comparison

### 3.2 Analysis datasets

Analysis populations:

- Intended to test (ITT): all samples intended to be tested
- Per protocol (PP): all samples with valid test results for the index test and reference standard

For the primary, diagnostic accuracy and time-to-result outcomes, the PP population will be analysed. For the feasibility endpoints, the ITT population will be analysed.

# 4 Description of statistical methods

## 4.1 Estimation of sensitivity and specificity

The following 2x2 table is defined:

Contingency table for analysis of diagnostic accuracy:

| RS | | | | |
|----|----------|----------|----------|-------|
| | | Positive | Negative | Total |
| IT | Positive | TP = a | FP = b | a+b |

| Negative | FN = c | TN = d | c+d |
|----------|--------|--------|---------|
| Total | a+c | b+d | a+b+c+d |

RS=reference standard, IT=index test, TP=true positive, FP=false positive, FN=false negative, TN=true negative

The diagnostic accuracy measures and their confidence intervals are estimated according to the following formulae:

Formulas and rules to calculate diagnostic accuracy measures:

| Measure | Formula | Confidence interval |
|-------------|---------|-----------------------------|
| Sensitivity | a/(a+c) | 2-sided 95%-Wilson-Score-CI |
| Specificity | d/(b+d) | 2-sided 95%-Wilson-Score-CI |

## 4.2 Analysis endpoints

 Estimates of sensitivity and specificity of Xpert MTB/XDR will be calculated compared to the reference standards defined below (for primary outcomes 1ad):

| DRUG RESISTANCE | COMPOSITE REFERENCE STANDARD |
|---|---|
| INH-resistant | NGS of $katG$ , $fabG1$ , $ahpC$ and $inhA$ detects $\geq 1$ mutation associated with INH resistance or MGIT culture is INH drug-resistant at the critical concentration. |
| ETH-resistant | NGS of <i>inhA</i> detects $\geq 1$ mutation associated with ETH resistance |
| FQ-resistant | NGS of $gyrA$ and $gyrB$ detects $\geq 1$ mutation associated with MFX resistance or MGIT culture is levofloxacin drug-resistant at the critical concentration. |
| Injectable-resistant | NGS of rrs, eis detects >1 mutation associated with injectable resistance or MGIT DST is kanamycin-resistant |
| INH-susceptible | NGS of <i>katG</i> , <i>fabG1</i> , <i>ahpC</i> and <i>inhA</i> does NOT detect any mutation associated with INH resistance and MGIT culture is INH-susceptible at the critical concentration. |
| ETH-susceptible | NGS of inhA does NOT detect any mutation associated with ETH resistance |
| FQ-susceptible | NGS of <i>gyrA</i> and <i>gyrB</i> does NOT detect any mutation associated with MFX resistance and MGIT culture is MFX-susceptible at the critical concentration. |
| Injectable-susceptible | NGS of <i>rrs</i> and <i>eis</i> does NOT detect any mutation associated with injectable-resistance and kanamycin MGIT DST is susceptible |

### Secondary outcomes:

- Estimates of sensitivity and specificity of Xpert MTB/XDR compared to WGS or phenotyping alone
- 2. Estimates of sensitivity and specificity of Xpert MTB/XDR to detect mutations in each gene target compared to WGS
- 3. Compare estimates of diagnostic accuracy of Xpert MTB/XDR to the estimates of diagnostic accuracy of SOC susceptibility testing against the composite reference standard using McNemar chi-square test
- Compare proportion of participants for whom valid susceptibility testing results become available based on Xpert MTB/XDR to the proportion of participants for whom valid susceptibility testing results become available based on SOC testing
- 5. Time-to-result comparing Xpert MTB/RIF Ultra testing to first results from Xpert MTB/XDR using Wilcoxon rank-sum test or t-test.
- 6. Feasibility
  - a. Proportion of participants with sufficient residual SR-sputum mix (≥2 ml) (total number of samples included as the denominator)
  - Median period between processing for Xpert MTB/RIF (preparation of SR-sputum mix) and the start of the Xpert MTB/XDR test
  - c. Determine the non-determinate rate of Xpert MTB/XDR (number of non-determinate result divided by total number of tests:
    - i. For each drug separately and combined for all
    - ii. Comparing specimens stored according to manufacturer recommendations (at 2-8°C for ≤4 hours or 25-35°C for ≤2.5 hours) and those exceeding those limits for operational reasons (Chisquared test)
    - iii. By Xpert MTB/RIF Ultra semi-quantitation result (chi-squared test)
    - iv. By sub-group (sufficient specimen, smear status, age group) (chi-squared test)
- 7. Exploratory analyses

## 5 Baseline descriptive statistics

Descriptive statistics tables will be generated to summarize the characteristics of the participants whose samples have been included in the study. The number of samples that have been included and excluded will be reported. Among the included participants, the information will be broken down by sex, age and ward type.

Results will be reported either in absolute numbers or summarized by mean, median, standard deviation, minimum, maximum and quartiles.

## 6 Planned interim analyses

No interim analyses are planned.

## 7 Additional sub-group analyses

Subgroups analyses are described in section 2.2 (6c iv and v)

Definition of sub-groups:

- Sufficient specimen: Group with ≥2 ml SR-sputum mix available vs. group with <2 ml SR-sputum mix
- Smear status: Positive for acid-fast bacilli (any quantitation) vs. negative for acid-fast bacilli
- Age group: Age <12 vs. age ≥12 years

# 8 Multiple comparisons/multiplicity adjustments

No multiple testing of statistical hypotheses will be performed.

## 9 Exploratory analyses

Exploratory analyses will be performed post hoc.

## 10 Sample size

A sample size of 320 specimens will be used in the diagnostic accuracy study. The sample size is dictated by the resources allocated to the project, and it is expected that the data generated will be combined in meta-analyses with other studies currently underway.

The sample size calculations detail the uncertainty of estimation of sensitivity among reference standard (RS)-positives and specificity among RS-negatives, expressed by the width of the 2-sided 95% confidence intervals. For technical reasons, the Pearson-Clopper-CI have been used in sample size considerations; the differences compared to the Wilson-Score-CI planned to be used in statistical analysis are negligible. The widths of the 95%-Pearson-Clopper-intervals for sensitivities / specificities of 70%, 80% or 90% were dependent on the expected prevalence of resistance to a specific anti-tuberculosis drugs (between 11 and 50%) and sample sizes of 320, 500 or 750. The width ranges from >30% (70% sensitivity at a prevalence [for RF-positive] of 11% among 320 patients) down to 4.7% (90% specificity at a prevalence [or RF-negative] of 89% among 750 patients).

The table shows expected prevalence of resistance to anti-tuberculosis drug class and the related number of resistant and susceptible specimens among 320, 500 and 750 participants together with confidence intervals for proportions of 70%, 80% and 90%:

| | | | | D+ or D- among | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Type of resistance | Resistant | Prev. | Measure | 320 | | | 500 | | | 750 | | |
| redistarioe | | | | N | ICL | uCL | N | ICL | uCL | N | ICL | uCL |
| | | 0.107 | n (Prev.) | 196 | | | 305 | | | 458 | | |
| | | | 70% Sens | 137 | 63.0% | 76.3% | 214 | 64.5% | 75.1% | 321 | 65.6% | 74.2% |
| | yes | 61% | 80% Sens | 157 | 73.7% | 85.4% | 244 | 75.1% | 84.3% | 366 | 76.0% | 83.6% |
| Isoniazid<br>resistance | | | 90% Sens | 176 | 84.9% | 93.8% | 275 | 86.1% | 93.1% | 412 | 86.9% | 92.6% |
| resistance | | | n (1-Prev.). | 125 | | | 195 | | | 293 | | |
| | | 200/ | 70% Spec | 88 | 61.2% | 77.9% | 137 | 63.0% | 76.3% | 205 | 64.4% | 75.2% |
| | no | 39% | 80% Spec | 100 | 71.9% | 86.6% | 156 | 73.7% | 85.4% | 234 | 75.0% | 84.4% |
| | | | 90% Spec | 113 | 83.4% | 94.6% | 176 | 84.9% | 93.8% | 264 | 86.0% | 93.2% |
| | | | n (Prev.) | 48 | | | 75 | | | 113 | | |
| | | 450/ | 70% Sens | 34 | 54.9% | 82.5% | 53 | 58.3% | 80.0% | 79 | 60.6% | 78.3% |
| | yes | 15% | 80% Sens | 38 | 65.9% | 90.2% | 60 | 69.2% | 88.4% | 90 | 71.4% | 86.9% |
| Second-line | | | 90% Sens | 43 | 77.6% | 96.9% | 68 | 80.9% | 95.7% | 102 | 82.9% | 94.9% |
| injectable<br>resistance | | | n (1-Prev.) | 272 | | | 425 | | | 638 | | |
| | | 85% | 70% Spec | 190 | 64.2% | 75.4% | 298 | 65.4% | 74.3% | 447 | 66.3% | 73.5% |
| | no | | 80% Spec | 218 | 74.7% | 84.6% | 340 | 75.9% | 83.7% | 510 | 76.7% | 83.0% |
| | | | 90% Spec | 245 | 85.8% | 93.3% | 383 | 86.7% | 92.7% | 574 | 87.4% | 92.2% |
| | | | n (Prev.) | 36 | | | 55 | | | 83 | | |
| | | | 70% Sens | 25 | 52.3% | 84.2% | 39 | 56.1% | 81.6% | 58 | 58.9% | 79.6% |
| | yes | 11% | 80% Sens | 29 | 63.2% | 91.5% | 44 | 67.0% | 89.6% | 66 | 69.8% | 88.0% |
| Fluoroquinolone | | | 90% Sens | 32 | 75.2% | 97.5% | 50 | 78.9% | 96.4% | 75 | 81.3% | 95.6% |
| resistance | | | n (1-Prev.). | 285 | | | 445 | | | 668 | | |
| | | 89% | 70% Spec | 200 | 64.3% | 75.3% | 312 | 65.5% | 74.2% | 468 | 66.4% | 73.5% |
| | no | | 80% Spec | 228 | 74.9% | 84.5% | 356 | 76.0% | 83.6% | 534 | 76.8% | 83.0% |
| | | | 90% Spec | 257 | 85.9% | 93.2% | 401 | 86.8% | 92.6% | 601 | 87.5% | 92.2% |
| | | | n (Prev.) | 160 | | | 250 | | | 375 | | |
| | | 500/ | 70% Sens | 112 | 62.3% | 77.0% | 175 | 63.9% | 75.6% | 263 | 65.1% | 74.6% |
| Ethionamide | yes | 50% | 80% Sens | 128 | 73.0% | 85.9% | 200 | 74.5% | 84.8% | 300 | 75.6% | 83.9% |
| | | | 90% Sens | 144 | 84.3% | 94.2% | 225 | 85.6% | 93.4% | 338 | 86.5% | 92.8% |
| resistance | | 500/ | n (1-Prev.) | 160 | | | 250 | | | 375 | | |
| | | | 70% Spec | 112 | 62.3% | 77.0% | 175 | 63.9% | 75.6% | 263 | 65.1% | 74.6% |
| | no | 50% | 80% Spec | 128 | 73.0% | 85.9% | 200 | 74.5% | 84.8% | 300 | 75.6% | 83.9% |
| | | | 90% Spec | 144 | 84.3% | 94.2% | 225 | 85.6% | 93.4% | 338 | 86.5% | 92.8% |

D+ =presence of resistance, D- =absence of resistance, Prev=prevalence, y=yes, n=no, ICL=lower confidence level, uCL=upper confidence level Red and green: widest and narrowest interval

Due to rounding errors, deviations of +/-1 case could occur for total N.

It is expected that a proportion of specimens will not be available for the diagnostic accuracy study because of an invalid Xpert MTB/XDR result, unavailability of a second or follow-up specimen and negative or contaminated culture. An additional 433 specimens will be required giving a final total of N=753:

Table: Number of specimens required to undergo Xpert MTB/XDR to achieve final sample size of N=320 for

diagnostic accuracy study, and anticipated enrolment period

| | UCT | | WHC | | Total |
|---|---|---|---|---|---|
| | % | N | % | N | N |
| Total specimens required | | 373 | | 380 | 753 |
| Available for feasibility study | 100 | 373 | 100 | 380 | 753 |
| Not available for diagnostic accuracy and time-to-result study | 41 | 153 | 71 | 280 | 433 |
| Insufficient specimen remaining for Xpert MTB/XDR | 1 | 4 | 1 | 4 | |
| Xpert MTB/XDR indeterminate | 5 | 19 | 5 | 19 | |
| No second / follow-up specimen | 10 | 37 | 40 | 152 | |
| Culture-negative or contaminated | 20 | 75 | 20 | 76 | |
| MGIT not available | 5 | 19 | 5 | 19 | |
| Available for diagnostic accuracy and time-to-result study | 59 | 220 | 29 | 100 | 320 |
| Enrolment period (@ 2 rifampicin-resistant specimens/day) | | 37 weeks | | 38 weeks | |

### 11 Minimization of error and bias

Consecutive, unselected samples with rifampicin-resistant MTB detected on Xpert Ultra testing in the routine laboratory will be used. These will include samples from a wide variety of facility types, geographical areas and patient/clinical backgrounds. Patients will only be excluded if they have been included previously, and not for any patient related factors. The study population will therefore be directly representative of the future target population and context of the Xpert MTB/XDR test.

Reference standard phenotyping, WGS and downstream bioinformatics analysis will be performed blinded to the index test result, which will have been performed in a different laboratory several weeks or months earlier.

## 11.1 Enrolment and randomization procedures

Enrolment will be consecutive rifampicin-resistant samples identified on routine Xpert MTB/RIF Ultra testing. There will be no randomisation.

### 12 Case definitions

The composite reference standard comprises phenotypic susceptibility testing and WGS performed on culture isolates. For the composite reference standard, samples will be defined as "resistant" if they are resistant by either phenotypic susceptibility testing or WGS and "susceptible" if they tested susceptible by both methods.

### 13 Statistical software

The analysis will be performed using Stata (version 16.1 or higher) and Microsoft Excel (version 2012).

# **14 References**

None

# **15 Document history**

| Version | Notes / Changes |
|---------|-------------------------------------------------|
| 1.0 | Initial version |
| 1.1 | Addressed comments by SO |
| 1.2 | Further corrections and removed tracked changes |